CLINICAL TRIAL: NCT04382144
Title: Levobupivacaine Versus Liposomal Bupivacaine (Exparel®) for Treatment of Pain and Disability in Lateral Epicondylitis - Off-Label, Investigator Initiated Randomized, Controlled, Double-Blind Cross-Over Treatment Trial
Brief Title: Levobupivacaine Versus Liposomal Bupivacaine (Exparel®) for Treatment of Pain and Disability in Lateral Epicondylitis
Acronym: LELIBU
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Markus Paakkonen, Head of Department, Hand Surgery, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TYKS/LeLiBu/1-2
Record Dates: First submitted 2020-04-28; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Tennis Elbow; Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: The trial will be a crossover study. During the pilot phase, we will recruit up to 6 patients, after which we will do a power analysis. In the main study, up to 25 patients will be randomized into 2 groups. Group 1 will receive an injection af levobupivacaine (Chirocaine) into the lateral epicondylitis. The outcomes are assessed over the next month and then they are given the injection of liposomal bupivacaine (Exparel).
  Normal distribution of data will be tested by Shapiro-Wilks test. The mean and Standard Deviation will be reported for normally distributed data. For data not distributed normally, the median and inter quartile ranges of the data will be reported.
  Independent samples t-test will be used for between-group comparison (normal distribution). The Mann-Whitney test will be used for non-normal data.
Who Masked: Care Provider
Masking Description: A nurse at the outpatient clinic will choose an envelope with the randomization information and assign the patient into their groups. The same nurse will prepare the injection, mask the syringe with a tape and give it to the doctor who will administer the injection. The same injection technique will be used for both drugs.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Levobupivacaine arm (Active Comparator): Patients will receive a single injection of 10 mL of 0.5% (5 mg/mL) levobupivacaine into the common extensor origin.
  Interventions: Drug: Liposomal bupivacaine
- Liposomal Bupivacaine arm (Experimental): Patients will receive a single injection of 10 mL (133mg) of liposomal bupivacaine into the common extensor origin.
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Patient will receive a single injection of a local anesthetic into the common extensor origin.

SUMMARY:
The main objective of the trial is to compare the effectiveness of injected levobupivacaine and liposomal bupivacaine in the treatment of pain and disability in patients with lateral epicondylitis.

Primary outcome is pain (VAS) at 1 week and at 1 month after injection. Secondary outcomes are the Quick Disabilities of the Arm, Shoulder and Hand DASH (Quick DASH) and Oxford Elbow Score (OES) and a record of time off work due to lateral epicondylitis in days at 1 week and at 1 month.

The study will be a cross-over trial

DETAILED DESCRIPTION:
This project compares bupivacaine and long acting liposomal bupivacaine in the treatment of pain and disability related to lateral epicondylitis.

The investigational medicinal products will be Chirocaine, ABBVIE OY, Espoo, Finland (levobupivacaine) and Exparel®, Pacira Pharmaceuticals, Inc., Parsippany, N.J. (liposomal bupivacaine).

The design of the study will be an off-label, investigator initiated, randomized, controlled, double-Blind cross over treatment trial. Exparel (liposomal bupivacaine) will be the medicinal product in the intervention arm, whilst Chirocaine (levobupivacaine) will serve as the active control.

Patients for the study will be recruited from the patients referred to the hand surgery outpatient clinic at Turku University Hospital, Finland.

During the pilot phase of the study, four patients will be recruited, after which power analysis is done. The main study will include up to 50 patients, 25 patients in each study arm. Patient enrollment will start immediately after the all the relevant permits have been obtained (estimated September 2020).

Normal distribution of data will be tested by Shapiro-Wilks test. The mean and Standard Deviation will be reported for normally distributed data. For data not distributed normally, the median and inter quartile ranges of the data will be reported. Independent samples t-test will be used for between-group comparison (normal distribution). The Mann-Whitney test will be used for non-normal data.

The results will be published in a peer reviewed international academic journal.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age 18-65
* employed
* chronic lateral epicondylitis (duration >3 months)
* pain in lateral epicondyle
* pain in resisted wrist extension in elbow extension (Cozen test)
* X-ray or Magnetic resonance imaging (MRI) of the elbow (<12 months from enrollment) with no pathological findings other than lateral epicondylitis

Exclusion Criteria:

* pregnancy, verbal confirmation from patient required
* unemployment
* allergy to levobupivacaine, bupivacaine or liposomal bupivacaine
* constant use of strong analgesics (e.g. opioids)
* other source of elbow pain (e.g. medial epicondylitis, distal biceps/triceps tendinitis)
* bilateral epicondylitis
* inability to give informed consent
* inability to understand the enrollment forms or to fill patient diary (forms are written in Finnish)
* previous injection treatment (e.g. cortisone, botulin toxin A, autologous plasma) for lateral epicondylitis during the past 3 months
* severe hepatic disease, or other underlying severe illness (cardiac failure, cancer, other systemic diseases)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain | 1 week
  pain at rest reported by patient on a Visual Analogue Scale (VAS), scale 0-100, higher value indicating worse outcome
Pain | 1 month
  pain at rest reported by patient on a Visual Analogue Scale (VAS), scale 0-100, higher value indicating worse outcome

SECONDARY OUTCOMES:
Pain | 1 week
  pain during grip reported by patient on Visual Analogue Scale (VAS),
Pain | 1 month
  pain during grip reported by patient on Visual Analogue Scale (VAS), scale 0-100, higher value indicating worse outcome
Disability | 1 week
  Patient reported outcome measure Disabilities of the Arm, Shoulder and Hand, scale 0-100, higher value indicating worse outcome
Disability | 1 month
  Patient reported outcome measure Disabilities of the Arm, Shoulder and Hand, scale 0-100, higher value indicating worse outcome
Disability | 1 week
  Patient reported outcome measure Oxford Elbow Score, scale 0-100, lower value indicating worse outcome
Disability | 1 month
  Patient reported outcome measure Oxford Elbow Score, scale 0-100, lower value indicating worse outcome
Disability | 1 week
  total number of days of work lost due to epicondylalgia
Disability | 1 month
  total number of days of work lost due to epicondylalgia
Pain | 1 week
  reduction in the amount of each pain medication taken
Pain | 1 month
  reduction in the amount of each pain medication taken

CONTACTS AND LOCATIONS:
Overall Officials: Markus Pääkkönen, PhD, Docent, Study Director — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No